CLINICAL TRIAL: NCT04667325
Title: Evaluation de l'Observance thérapeutique à la spirométrie Incitative Chez Les Patients drépanocytaires
Brief Title: Evaluation of Therapeutic Adherence to Inciting Spirometry in Sickle Cell Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: KINEDREP
Record Dates: First submitted 2020-11-30; First posted 2020-12-14 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Sickle Cell Disease
Keywords: acute chest syndrome, incentive spirometry, compliance
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sickle cell disease is one of the most common genetic diseases in the world. (1) It is characterized by the production of abnormal hemoglobin mainly responsible for vaso-occlusive clinical manifestations and chronic hemolysis with anemia. (2) It is therefore a chronic disease with major acute complications, such as acute chest syndrome. The treatment for this syndrome will be based on oxygenation, hydration and analgesia. At the physiotherapy level, we will have an action on the prevention and treatment of the syndrome by incentive spirometry. (3,4) In fact, it is currently the only physiotherapy treatment that has proven its effectiveness and is recommended for sickle cell patients. (3) As part of prevention, it is recommended to prescribe incentive spirometry during vaso-occlusive crisis. It has been shown to reduce the risk of atelectasis and significantly limit the risk of developing ACS. (5) In treatment, it makes it possible to regain normal chest amplification and therefore to allow ventilation of unventilated areas. (3.4) However, in order to increase therapeutic efficacy, patient compliance is essential.

Adherence to treatment is a major problem in chronic diseases. Currently, it is estimated that 80% of patients with chronic conditions do not sufficiently follow their therapy, which limits the optimization of benefits. (6) This is the case in sickle cell patients, especially with hydroxyurea which is their disease-modifying treatment. Lack of adherence is the most common cause of primary failure of this treatment.

During various treatments, we noticed the patients' lack of compliance with spirometry. Indeed, we explained to the patient how to do the incentive spirometry, so that he could practice it several times a day as recommended. When we returned the next day, or after a weekend, most of the time the patients had little or no observance. So I wanted to know if this concerns a majority of patients with sickle cell disease. Indeed, it appears important to assess compliance in these patients in order to improve the effectiveness of treatment and reduce the risk of ACS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease,
* Major
* No opposition for participation in the protocol

Exclusion Criteria:

* Patients unable to answer the questionnaire due to linguistic or other problems
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with sickle cell anemia
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
To take stock of the observance of sickle cell patients with inciting spirometry | Through study completion, an everage of 10 minutes
  Measuring compliance through the questionnaire

SECONDARY OUTCOMES:
To take stock of patients' knowledge of their pathology and incentive spirometry | Through study completion, an everage of 10 minutes
  Assessing knowledge about their pathology and treatment via the questionnaire
Measuring adherence to medical follow-up | Through study completion, an everage of 10 minutes
  Measuring the number of consultations via the questionnaire
Assessing the impact of the disease on quality of life | Through study completion, an everage of 10 minutes
  Measuring the patient's quality of life via the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier intercommunal de Créteil, Créteil, France